CLINICAL TRIAL: NCT00801489
Title: A Phase 2 Study of Fludarabine, Cytarabine, Filgrastim-sndz,Gemtuzumab Ozogamicin and Idarubicin in Newly Diagnosed Core Binding Factor Associated Acute Myelogenous Leukemia
Brief Title: Fludarabine Phosphate, Cytarabine, Filgrastim-sndz, Gemtuzumab Ozogamicin, and Idarubicin Hydrochloride in Treating Patients With Newly Diagnosed Acute Myeloid Leukemia or High-Risk Myelodysplastic Syndrome
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Collaborators: National Cancer Institute (NCI) (NIH)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2007-0147; NCI-2012-01659 (Registry Identifier: CTRP (Clinical Trial Reporting Program)); 2007-0147 (Other: M D Anderson Cancer Center)
Record Dates: First submitted 2008-12-02; First posted 2008-12-03 (Estimated); Last update posted 2025-10-09 (Actual); Status verified 2025-10

CONDITIONS: Acute Myeloid Leukemia With Inv(16)(p13.1q22); CBFB-MYH11; Acute Myeloid Leukemia With t(16;16)(p13.1;q22); CBFB-MYH11; Acute Myeloid Leukemia With t(8;21); (q22; q22.1); RUNX1-RUNX1T1; de Novo Myelodysplastic Syndrome; High Risk Myelodysplastic Syndrome; Inv(16); Myelodysplastic Syndrome With Excess Blasts; t(16;16); t(8;21); Untreated Adult Acute Myeloid Leukemia
MeSH Terms: conditions — Leukemia, Myelomonocytic, Acute; Anemia, Refractory, with Excess of Blasts | interventions — Cytarabine; Decitabine; Injections; Filgrastim; Granulocyte Colony-Stimulating Factor; fludarabine phosphate; Gemtuzumab; Idarubicin

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: Yes | FDA-regulated Device: No

ARMS (1):
- Treatment (filgrastim, fludara, cytara, gemtuzu, idarubicin) (Experimental): See Detailed Description
  Interventions: Drug: Cytarabine; Drug: Decitabine; Biological: Filgrastim-sndz; Drug: Fludarabine Phosphate; Drug: Gemtuzumab Ozogamicin; Drug: Idarubicin; Other: Laboratory Biomarker Analysis

INTERVENTIONS:
Drug: Cytarabine — Given IV
  Other Names: .beta.-Cytosine arabinoside; 1-.beta.-D-Arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-.beta.-D-Arabinofuranosylcytosine; 1-Beta-D-arabinofuranosyl-4-amino-2(1H)pyrimidinone; 1-Beta-D-arabinofuranosylcytosine; 1.beta.-D-Arabinofuranosylcytosine; 2(1H)-Pyrimidinone, 4-Amino-1-beta-D-arabinofuranosyl-; 2(1H)-Pyrimidinone, 4-amino-1.beta.-D-arabinofuranosyl-; Alexan; Ara-C; ARA-cell; Arabine; Arabinofuranosylcytosine; Arabinosylcytosine; Aracytidine; Aracytin; Aracytine; Beta-cytosine Arabinoside; CHX-3311; Cytarabinum; Cytarbel; Cytosar; Cytosine Arabinoside; Cytosine-.beta.-arabinoside; Cytosine-beta-arabinoside; Erpalfa; Starasid; Tarabine PFS; U 19920; U-19920; Udicil; WR-28453
Drug: Decitabine — Given IV
  Other Names: 5-Aza-2'-deoxycytidine; Aza-TdC; Dacogen; Decitabine for Injection; Deoxyazacytidine; Dezocitidine
Biological: Filgrastim-sndz — Given SC
  Other Names: Filgrastim Biosimilar Filgrastim-sndz; Zarxio
Drug: Fludarabine Phosphate — Given IV
  Other Names: 2-F-ara-AMP; 9H-Purin-6-amine, 2-fluoro-9-(5-O-phosphono-.beta.-D-arabinofuranosyl)-; Beneflur; Fludara; SH T 586
Drug: Gemtuzumab Ozogamicin — Given IV
  Other Names: Calicheamicin-Conjugated Humanized Anti-CD33 Monoclonal Antibody; CDP-771; CMA-676; gemtuzumab; hP67.6-Calicheamicin; Mylotarg; WAY-CMA-676
Drug: Idarubicin — Given IV
  Other Names: 4-Demethoxydaunomycin; 4-demethoxydaunorubicin; 4-DMDR
Other: Laboratory Biomarker Analysis — Correlative studies

SUMMARY:
This phase II trial studies the side effects and how well fludarabine phosphate, cytarabine, filgrastim-sndz, gemtuzumab ozogamicin, and idarubicin hydrochloride work in treating patients with newly diagnosed acute myeloid leukemia or high-risk myelodysplastic syndrome. Drugs used in chemotherapy, such as fludarabine phosphate, cytarabine, and idarubicin hydrochloride, work in different ways to stop the growth of cancer cells, either by killing the cells or by stopping them from dividing. Gemtuzumab ozogamicin is a monoclonal antibody, called gemtuzumab, linked to a antitumor drug, called calicheamicin. Gemtuzumab is a form of targeted therapy because it attaches to specific molecules (receptors) on the surface of cancer cells, known as CD33 receptors, and delivers calicheamicin to kill them. Colony-stimulating factors, such as filgrastim-sndz, may increase the number of immune cells found in bone marrow or peripheral blood and may help the immune system recover from the side effects of chemotherapy. Giving fludarabine phosphate, cytarabine, filgrastim-sndz, gemtuzumab ozogamicin, and idarubicin hydrochloride may kill more cancer cells.

DETAILED DESCRIPTION:
PRIMARY OBJECTIVES:

I. Evaluate the safety of a regimen incorporating fludarabine phosphate (fludarabine), high-dose cytarabine, filgrastim-sndz, gemtuzumab ozogamicin and idarubicin hydrochloride (idarubicin) in patients with untreated inv(16) or t(8;21) acute myeloid leukemia (AML).

II. Evaluate the complete remission rates achieved in this population with this regimen.

SECONDARY OBJECTIVES:

I. Assess the proportion of patients with untreated inv(16) or t(8;21) AML who, having entered complete remission (CR) on this regimen, remain alive in CR two years from CR date.

II. Assess whether the quantitative polymerase chain reaction (Q-PCR) results can be used in detecting relapse in these patients.

OUTLINE:

REMISSION INDUCTION: Patients receive filgrastim-sndz subcutaneously (SC) once daily (QD) beginning on day -1 and continuing until blood count recovery. Patients also receive fludarabine phosphate intravenously (IV) over 30 minutes on days 1-5, cytarabine IV over 4 hours on days 1-5, gemtuzumab ozogamicin IV over 2 hours on day 1. Patients not in remission after their first induction therapy may repeat remission induction therapy.

POST-REMISSION THERAPY: Patients receive filgrastim-sndz SC on day -1, fludarabine phosphate IV over 30 minutes on days 1-3, cytarabine IV over 4 hours on days 1-3, gemtuzumab ozogamicin IV over 2 hours on day 1 of courses 1 or 2 and 5 or 6, and idarubicin hydrochloride IV over 30 minutes on days 2 and 3 of one post-remission course (post-remission courses 3 or 4) determined by the treating physician after discussion with the PI if suboptimal qPCR response (qPCR > 0.01 after post-remission cycle 2 or 3). Treatment repeats every 4-6 weeks for up to 6 courses in the absence of disease progression or unacceptable toxicity.

FURTHER MODIFICATION OF POST-REMISSION THERAPY: Patients older than 60, with significant comorbidities, experiencing life-threatening complications, prolonged cytopenias, or not achieving complete molecular response may receive decitabine IV over 1 hour daily for 5 days after discussion with the principal investigator. Treatment repeats every 4-6 weeks for up to 12 courses in the absence of disease progression or unacceptable toxicity.

After completion of study treatment, patients are followed up every 6 months for 2 years.

ELIGIBILITY:
Inclusion Criteria:

* Patients must have untreated AML, or high-risk myelodysplastic syndromes (MDS) (refractory anemia with excess blasts, [RAEB], or RAEB "in transformation" [RAEB-t]) characterized by t(8;21), inv(16), or t(16;16); the presence of additional abnormalities is irrelevant
* Patients must provide written consent
* Participants will not be excluded based on performance status; for patients with Eastern Cooperative Oncology Group (ECOG) performance status >= to 3 the dosing schedule will be discussed with study chairman
* Patients with organ dysfunction will not be excluded from the study; for patients with evidence of organ dysfunction (creatinine >= 1.5, cardiac ejection fraction =< 50%, total bilirubin >=2 and aspartate aminotransferase [AST]/alanine aminotransferase [ALT] >= 3 times upper limit of normal [ULN]), dose adjustments/omissions will be made
* Up to one cycle of prior induction therapy will be permitted to include patients in whom presence of "good-risk" cytogenetics was initially missed; if the patient is in remission from induction therapy, he/she will receive post-remission therapy; if the patient is not in remission then he/she will receive induction therapy
* Patients of child bearing potential should practice effective methods of contraception

Exclusion Criteria:

* Pregnant and lactating females will be excluded

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 270 (Estimated)
Dates: Start 2007-04-04 (Actual); Primary Completion 2028-10-11 (Estimated); Study Completion 2028-10-11 (Estimated)

PRIMARY OUTCOMES:
Complete remission rate | Up to 2 years
Toxicity rate | Up to 2 years

CONTACTS AND LOCATIONS:
Overall Officials: Gautam Borthakur, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- M D Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- See also: MD Anderson Cancer Center — http://www.mdanderson.org